CLINICAL TRIAL: NCT03101748
Title: A Phase 1b Study of Neratinib, Pertuzumab, and Trastuzumab With Taxol (3HT) in Metastatic and Locally Advanced Breast Cancer, and Phase II Study of 3HT Followed by AC in HER2 + Primary IBC, and Neratinib With Taxol (NT) Followed by AC in HR+ /HER2- Primary IBC
Brief Title: Neratinib and Paclitaxel With or Without Pertuzumab and Trastuzumab Before Combination Chemotherapy in Treating Patients With Metastatic or Locally Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: <75% accrued
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0537; NCI-2017-00813 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0537 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Breast Inflammatory Carcinoma; Locally Advanced Breast Carcinoma; Metastatic Breast Carcinoma; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; neratinib; Paclitaxel; Taxes; pertuzumab; 2C4 antibody; Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Cohort 1 Phase Ib) (Experimental): Patients receive neratinib PO QD on days 1-21, paclitaxel IV over 1-3 hours on days 1, 8, and 15, pertuzumab IV over 1 hour on day 1, and trastuzumab IV over 1-2 hours on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients without progression or excessive toxicity with metastatic disease may receive up to 4 additional courses and with locally advanced disease may receive up to 2 additional courses.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Neratinib; Drug: Paclitaxel; Biological: Pertuzumab; Biological: Trastuzumab
- Group B (Cohort 1 Phase II) (Experimental): Patients receive neratinib, paclitaxel, pertuzumab, and trastuzumab as in Group A. Patients then receive doxorubicin IV and cyclophosphamide IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Other: Laboratory Biomarker Analysis; Drug: Neratinib; Drug: Paclitaxel; Biological: Pertuzumab; Biological: Trastuzumab
- Group C (Cohort 2) (Experimental): Patients receive neratinib PO QD on days 1-21, paclitaxel IV over 1-3 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery/ Patients then receive doxorubicin and cyclophosphamide as in Group B. Patients then undergo standard of care surgery.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Other: Laboratory Biomarker Analysis; Drug: Neratinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Group B (Cohort 1 Phase II); Group C (Cohort 2)
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
  Arms: Group B (Cohort 1 Phase II); Group C (Cohort 2)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Neratinib — Given PO
  Other Names: (2E)-N-(4-((3-chloro-4-((pyridin-2-yl)methoxy)phenyl)amino)-3-cyano-7-ethoxyquinolin-6-yl)-4-(dimethylamino)but-2-enamide; HKI 272; HKI-272; PB 272; PB-272
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pertuzumab — Given IV
  Other Names: 2C4; 2C4 Antibody; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; rhuMAb2C4; RO4368451
  Arms: Group A (Cohort 1 Phase Ib); Group B (Cohort 1 Phase II)
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
  Arms: Group A (Cohort 1 Phase Ib); Group B (Cohort 1 Phase II)

SUMMARY:
This phase I/II trial studies the side effect and best dose of neratinib and to see how well it works with paclitaxel and with or without pertuzumab and trastuzumab before combination chemotherapy in treating patients with breast cancer that has spread to other places in the body (metastatic). Neratinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with pertuzumab and trastuzumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as paclitaxel, doxorubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving neratinib, pertuzumab, trastuzumab, paclitaxel and combination chemotherapy may work better in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of neratinib in combination with paclitaxel, pertuzumab, and trastuzumab in HER2-positive (HER2+) metastatic or locally advanced (stage III) breast cancer within 2 cycles. (Cohort 1: Phase Ib) II. To determine the pathologic complete response (pCR) rate of neratinib in combination with paclitaxel, pertuzumab, and trastuzumab followed by doxorubicin and cyclophosphamide (AC) in HER2+ metastatic or locally advanced (stage III) inflammatory breast cancer (IBC) patients. (Cohort 1: Phase II) III. To determine the pCR rate of neratinib in combination with paclitaxel followed by AC in HER2-negative/hormone receptor (HR)-positive (HER2-/HR+) metastatic or locally advanced (stage III) IBC patients. (Cohort 2)

SECONDARY OBJECTIVES:

I. To estimate 2 years progression free survival (PFS) rate of HER2+ metastatic or locally advanced (stage III) IBC patients, and HER2-/HR+ IBC patients treated with neratinib plus anthracycline and taxane based chemotherapy. (Cohort I Phase II and Cohort II) II. To determine toxicity and safety of the combination therapy.

EXPLORATORY OBJECTIVES:

I. To determine the adaptive target and downstream changes in pan-HER family members induced by one-week window period of neratinib based on tissue and blood based biomarkers.

II. To determine the correlation between positive/negative changes in EGFR, HER2 and HER4 and the occurrence of pCR.

III. To determine the rate of HER2 mutation in HER2+ IBC and HER2-/HR+ IBC. IV. To determine the association between HER2 mutation and pCR achieved by study combination therapy.

V. To determine the correlation between tumor tissue based pharmacodynamic marker changes in association with circulating tumor cells (CTC) and circulating tumor deoxyribonucleic acid (ctDNA).

OUTLINE: This is a phase I, dose-escalation study of neratinib followed by a phase II study. Patients are assigned to 1 of 3 groups.

GROUP A (COHORT 1 PHASE IB): Patients receive neratinib orally (PO) once daily (QD) on days 1-21, paclitaxel intravenously (IV) over 1-3 hours on days 1, 8, and 15, pertuzumab IV over 1 hour on day 1, and trastuzumab IV over 1-2 hours on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients without progression or excessive toxicity with metastatic disease may receive up to 4 additional courses and with locally advanced disease may receive up to 2 additional courses.

GROUP B (COHORT 1 PHASE II): Patients receive neratinib, paclitaxel, pertuzumab, and trastuzumab as in Group A. Patients then receive doxorubicin IV and cyclophosphamide IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgery.

GROUP C (COHORT 2): Patients receive neratinib PO QD on days 1-21, paclitaxel IV over 1-3 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery/ Patients then receive doxorubicin and cyclophosphamide as in Group B. Patients then undergo standard of care surgery.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast cancer
* Able to provide written informed consent for the trial
* Performance status of =< 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Able to swallow oral medication
* Left ventricular ejection fraction (LVEF) assessment by 2-dimensional (D) echocardiogram or multi-gated acquisition (MUGA) scan performed within 90 days prior to registration must be >= 50%
* Absolute neutrophil count >= 1,500 /uL
* Platelets >= 100,000 /uL
* Hemoglobin >= 9 g/dL
* Creatinine clearance >= 50 ml/min
* Total bilirubin =< 1.5 X upper limit of normal (ULN), for patients with congenital unconjugated hyperbilirubinemia (Crigler-Najjar syndrome type 1 and 2, Gilbert syndrome) that transient hyperbilirubinemia can occur due to physiological condition, as long as there is clear documentation of diagnosis, allowed to be enrolled if direct (conjugated) bilirubin is =< 1.5 X ULN
* Alanine aminotransferase and aspartate aminotransferase =< 2.5 X ULN except in patients with aspartate aminotransferase (AST)/alanine aminotransferase (ALT) elevation that is declared to be caused due to liver metastasis, they are allowed to be enrolled as long as < 5 x ULN
* Subject of childbearing potential should be willing to use effective methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study and through at least 4 months after the last dose of study drug; subject of childbearing potential is defined as has not been surgically sterilized or free from menses for > 1 year; effective methods of birth control include: 1) use of hormonal birth control methods: pills, shots/injections, implants (placed under the skin by a health care provider), or patches (placed on the skin); 2) intrauterine devices (IUDs); 3) using 2 barrier methods (each partner must use 1 barrier method) with a spermicide; males must use the male condom (latex or other synthetic material) with spermicide; females must choose either a diaphragm with spermicide, or cervical cap with spermicide, or a sponge (spermicide is already in the contraceptive sponge); female patients of childbearing potential must have a negative urine pregnancy test no more than 7 days prior to starting study drug; 4) for male participant, they must agree and commit to use a barrier method of contraception while on treatment and for 3 months after the last dose of investigational product
* Cohort 1: Phase 1b: patient must have HER2 + (regardless of hormonal receptor status) metastatic or locally advanced breast cancer (IBC or Non-IBC); HER2 positive status is defined as strongly positive (3+) staining score by immunohistochemistry (IHC), or gene amplification using fluorescence in situ hybridization (FISH), if performed; if IHC is equivocal (2+), please refer to current American Society of Clinical Oncology (ASCO) guidelines algorithm for evaluation of HER2; HER2 negative status, which is determined by assays using IHC require negative (0 or 1+) staining score; if IHC is equivocal (2+) staining score, please refer to current ASCO guidelines algorithm for evaluation of HER2; IBC is determined by using international consensus criteria: onset: rapid onset of breast erythema, edema and/or peau d'orange, and/or warm breast, with/without an underlying breast mass; duration: history of such findings no more than 6 months; extent erythema occupying at least 1/3 of whole breast; pathology: pathologic confirmation of invasive carcinoma
* Cohort 1: Phase II: patient must have HER2+ (regardless of hormonal receptor status) stage III IBC or Stage IV IBC if the metastatic sites are amenable for local therapy (i.e. radiation and/ or surgery) and will have breast surgery
* Cohort 2: Patient must have HER2-/HR+ stage III IBC or Stage IV IBC if the metastatic sites are amenable for local therapy (i.e. radiation and/ or surgery) and will have breast surgery

Exclusion Criteria:

* Excisional biopsy or lumpectomy for the current breast cancer
* Any other previous malignancies (except for cervical in situ cancers treated only by local excision, and basal and squamous cell carcinomas of the skin) within 5 years
* Any other previous antitumor therapies for the current cancer event; this exclusion does not apply to phase Ib part of cohort 1
* Breast-feeding at screening or planning to become pregnant during the course of therapy
* History of active or known autoimmune disease that can cause diarrhea like (but not limited to) Addison's disease, celiac disease/gluten intolerance/irritable bowel syndrome, scleroderma
* Active infection or chronic infection requiring chronic suppressive antibiotics
* Known hepatitis B or hepatitis C with abnormal liver function tests
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function
* Persistent >= grade 2 diarrhea regardless of etiology
* Sensory or motor neuropathy >= grade 2
* Conditions that would prohibit intermittent administration of corticosteroids for paclitaxel premedication; however, corticosteroid can be dropped after confirming of no asthma like reaction to paclitaxel after 3 doses
* Uncontrolled hypertension defined as a systolic blood pressure (BP) > 150 mmHg or diastolic BP > 90 mmHg, with or without anti-hypertensive medications
* Cardiac disease (history of and/or active disease) that would preclude the use of any of the drugs included in the treatment regimen; this includes but is not confined to:

  * Active cardiac diseases including:

    * Symptomatic angina pectoris within the past 180 days that required the initiation of or increase in anti-anginal medication or other intervention
    * Ventricular arrhythmias except for benign premature ventricular contractions
    * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
    * Conduction abnormality requiring a pacemaker
    * Valvular disease with documented compromise in cardiac function
    * Symptomatic pericarditis
  * History of cardiac disease:

    * Myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function
    * History of documented congestive heart failure (CHF)
    * Documented cardiomyopathy
* If you are pregnant, you will not be enrolled on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Layman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lim B, Marx A, Kai M, Alexander A, Bassett R Jr, Ma W, Willey J, Sun H, Nasrazadani A, Mohammad MM, Zhang J, Lucci A, Sun SX, Stauder MC, Whitman GJ, Le-Petross H, Valero V; MDACC Inflammatory Breast Cancer Team; Woodward WA, Layman RM. A phase Ib/II trial of neoadjuvant neratinib added to standard therapy in patients with HER2-positive or HR-positive/HER2-negative inflammatory breast cancer (including stage III and IV disease). Ther Adv Med Oncol. 2025 Oct 14;17:17588359251379392. doi: 10.1177/17588359251379392. eCollection 2025. PMID 41116969
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Feb 2018~ Oct 2021. All recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: 43 patients were accrued and assessed for eligibility and 34 patients were assigned to the cohort.
Groups:
- Cohort 1 Phase Ib Dose Level -1: HER2-positive breast cancer patients received neratinib 40 mg daily in combination with paclitaxel, pertuzumab, and trastuzumab.
- Cohort 1 Phase Ib Dose Level 0: HER2-positive breast cancer patients received neratinib 80 mg daily in combination with paclitaxel, pertuzumab, and trastuzumab.
- Cohort 1 Phase Ib Dose Level 1: HER2-positive breast cancer patients received neratinib 120 mg daily in combination with paclitaxel, pertuzumab, and trastuzumab.
- Cohort 1 Phase Ib Dose Level 2: HER2-positive breast cancer patients received neratinib 160 mg daily in combination with paclitaxel, pertuzumab, and trastuzumab.
- Cohort 1 Phase Ib Dose Level 3: HER2-positive breast cancer patients received neratinib 200 mg daily in combination with paclitaxel, pertuzumab, and trastuzumab.
- Cohort 1 Phase II: HER2-positive inflammatory breast cancer patients received neratinib at the recommended Phase II dose (RP2D) in combination with paclitaxel, pertuzumab, and trastuzumab, followed by doxorubicin and cyclophosphamide.
- Cohort 2: HER2-negative, hormone receptor-positive inflammatory breast cancer patients received neratinib 200 mg daily in combination with paclitaxel, followed by doxorubicin and cyclophosphamide.
Period: Overall Study
Arm/Group | Cohort 1 Phase Ib Dose Level -1 | Cohort 1 Phase Ib Dose Level 0 | Cohort 1 Phase Ib Dose Level 1 | Cohort 1 Phase Ib Dose Level 2 | Cohort 1 Phase Ib Dose Level 3 | Cohort 1 Phase II | Cohort 2
Started | 0 | 2 | 2 | 0 | 0 | 14 | 16
Completed | 0 | 1 | 1 | 0 | 0 | 9 | 10
Not Completed | 0 | 1 | 1 | 0 | 0 | 5 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 1 | 0 | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: No participants enrolled on Cohort 1 Phase Ib Dose Level -1, Cohort 1 Phase Ib Dose Level 2, or Cohort 1 Phase Ib Dose Level 3
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Phase Ib Dose Level -1 | Cohort 1 Phase Ib Dose Level 0 | Cohort 1 Phase Ib Dose Level 1 | Cohort 1 Phase Ib Dose Level 2 | Cohort 1 Phase Ib Dose Level 3 | Cohort 1 Phase II | Cohort 2 | Total
Number analyzed (Participants) | 0 | 2 | 2 | 0 | 0 | 14 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2 | 0 | 0 | 12 | 16 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 2 |  |  | 14 | 16 | 34
  Male |  | 0 | 0 |  |  | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0 |  |  | 4 | 2 | 6
  Not Hispanic or Latino |  | 2 | 2 |  |  | 10 | 13 | 27
  Unknown or Not Reported |  | 0 | 0 |  |  | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0 |  |  | 1 | 0 | 1
  Asian |  | 1 | 0 |  |  | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander |  | 0 | 0 |  |  | 0 | 0 | 0
  Black or African American |  | 0 | 0 |  |  | 1 | 2 | 3
  White |  | 1 | 2 |  |  | 12 | 11 | 26
  More than one race |  | 0 | 0 |  |  | 0 | 2 | 2
  Unknown or Not Reported |  | 0 | 0 |  |  | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2 |  |  | 14 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Dose-Limiting Toxicities (DLTs) During Dose Escalation
Description: Dose-limiting toxicities (DLTs) observed during the first two treatment cycles (approximately 6 weeks) among participants receiving escalating doses of neratinib in combination therapy in Cohort I Phase Ib. Participants With ≥1 DLT.
Time Frame: From treatment initiation through completion of 2 cycles (approximately 6 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Phase Ib Dose Level -1 | Cohort 1 Phase Ib Dose Level 0 | Cohort 1 Phase Ib Dose Level 1 | Cohort 1 Phase Ib Dose Level 2 | Cohort 1 Phase Ib Dose Level 3
Number analyzed (Participants) | 0 | 2 | 2 | 0 | 0
Participants |  | 0 | 2 |  |

2. Primary Outcome: Pathologic Complete Response (pCR) in HER2+ Metastatic or Locally Advanced IBC in Cohort I Phase II
Description: Pathologic complete response (pCR) was defined as no residual invasive cancer in the breast and sampled lymph nodes at surgery (ypT0/Tis, ypN0). The primary analysis was conducted using the intent-to-treat (ITT) population; participants who did not undergo surgery were counted as non-pCR.
Time Frame: At surgery following completion of neoadjuvant therapy (approximately 18-24 weeks from treatment initiation).
Population: All patients who initiated protocol treatment were included in the intent-to-treat (ITT) population in Cohort I Phase II.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 Phase II
Number analyzed (Participants) | 14
Participants | 5

3. Primary Outcome: Pathologic Complete Response (pCR) in HER2-Negative / HR-Positive IBC in Cohort II
Description: as for outcome 2
Time Frame: At the time of surgery (mastectomy), following completion of neoadjuvant therapy; approximately 18-24 weeks from treatment initiation.
Population: All patients who initiated protocol treatment were included in the intent-to-treat (ITT) population in Cohort II.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort II: HER2-negative, hormone receptor-positive inflammatory breast cancer patients received neratinib 200 mg daily in combination with paclitaxel, followed by doxorubicin and cyclophosphamide.
Arm/Group | Cohort II
Number analyzed (Participants) | 16
Participants | 1

4. Secondary Outcome: Event-Free Survival (EFS) Rate at 2 Years
Description: Event-free survival (EFS) was defined as the time from treatment initiation to the first occurrence of disease progression, recurrence, or death from any cause. EFS rates at 2 years were estimated using the Kaplan-Meier method; participants without an event were censored at last disease assessment.
Time Frame: From treatment initiation to 2 years after start of therapy.
Population: All patients who initiated protocol treatment were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 Phase II | Cohort 2
Number analyzed (Participants) | 14 | 16
percentage of participants | 84.6 [67.1 to 100] | 68.2 [48.6 to 95.7]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed for 2 years after treatment discontinuation, up to 3 years; all Adverse Events were collected from the time of the first protocol-specific intervention until 30 days after the last dose of drug, up to 1 year
Description: Adverse events were assessed using CTCAE v4.0. All AEs of ≥ Grade 2 for non-hematologic events and ≥ Grade 3 for hematologic events, regardless of attribution, were recorded.
Arm/Group | Cohort 1 Phase Ib Dose Level 0 | Cohort 1 Phase Ib Dose Level 1 | Cohort 1 Phase II | Cohort 2
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/2 | 2/14 | 5/16
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 6/14 | 3/16
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 14/14 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Phase Ib Dose Level 0 (N=2) | Cohort 1 Phase Ib Dose Level 1 (N=2) | Cohort 1 Phase II (N=14) | Cohort 2 (N=16)
Fever (General disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Urinary tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Edema limbs (General disorders) | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Breast Infection (Infections and infestations) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
BUN Increased " (Investigations) | 0 | 0 | 1 | 0
Creatinine Increased (Renal and urinary disorders) | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urine output decreased (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Stone (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 Phase Ib Dose Level 0 (N=2) | Cohort 1 Phase Ib Dose Level 1 (N=2) | Cohort 1 Phase II (N=14) | Cohort 2 (N=16)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 14 | 14
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0
Breast Infection (Infections and infestations) | 0 | 0 | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Concentration Impairment (Nervous system disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 14 | 15
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 3 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1 | 0
Syte (Eye disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 9 | 8
Fever (General disorders) | 0 | 1 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 3 | 2
Hypertension (Vascular disorders) | 1 | 0 | 3 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
COVID-19 or SARS-CoV-2 infection (Infections and infestations) | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 0 | 1
Lung Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0
Mucositis Oral (Gastrointestinal disorders) | 1 | 1 | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nail Infection (Infections and infestations) | 0 | 1 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 13 | 7
Neutrophil count decreased (Investigations) | 0 | 1 | 2 | 2
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Paresthesia (Nervous system disorders) | 1 | 1 | 3 | 2
Paronychia (Infections and infestations) | 2 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Vascular disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 7 | 5
Renal calculi (Renal and urinary disorders) | 0 | 0 | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 0 | 3 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 3 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 2 | 3
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 5 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 0
Vaginal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Vaginal Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 8 | 4
Weight gain (Investigations) | 0 | 1 | 0 | 2
Weight loss (Investigations) | 0 | 0 | 4 | 4
White blood cell decreased (Investigations) | 0 | 1 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03101748/Prot_SAP_001.pdf
  • Informed Consent Form (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/48/NCT03101748/ICF_000.pdf